#### **PROTOCOL**

STUDY TITLE:

Investigation of Ranibizumab for the Treatment

of Persistent Diabetic Neovascularization as

Assessed by Super Wide-Field Angiography

(Optos)

STUDY DRUG

Recombinant humanized anti-VEGF

monoclonal antibody fragment (rhuFab V2

[ranibizumab])

**SPONSOR** 

Rush University Medical Center

1725 West Harrison, Suite 915, Chicago, IL 60612

Phone: 312-942-2117

Fax: 312-563-2607

IND:

**INVESTIGATOR** 

Mathew W. MacCumber, MD, PhD

SUB-

Jack Cohen, MD

**INVESTIGATORS** 

Michael J. Davis, MD Pauline Merrill, MD

Kirk Packo, MD

**DATE FINAL:** 

28 DEC 06

ORA#: 06120402

IRB APPROVAL DATE: 8/15/07 IRB EXPIRATION DATE: 8/15/08

## **TABLE OF CONTENTS**

| | | | Page |
|----|------|-----------------------------------------|------|
| 1. | BAC | KGROUND | 1 |
| | 1.1 | Pathophysiology | 1 |
| | 1.2 | Treatment | 1 |
| | 1.3 | Ranibizumab | 1 |
| | 1.4 | Nonclinical Experience with Ranibizumab | 1 |
| | | 1.4.1 Nonclinical Pharmacokinetics | 1 |
| | | 1.4.2 Nonclinical Toxicology | 2 |
| | | 1.4.3 Stability Studies | 2 |
| | 1.5 | Clinical Experience with Ranibizumab | 2 |
| | | 1.5.1 Study FVF1770g | 2 |
| | | 1.5.2 Study FVF2128g | 3 |
| | | 1.5.3 Study FVF2425g. | 3 |
| | | 1.5.4 Study FVF2428g. | 3 |
| | | 1.5.5 Study FVF2508g | 3 |
| | | 1.5.6 Study FVF2587g | 4 |
| | | 1.5.7 Study FVF2598g | 4 |
| | | 1.5.8 Study FVF3192g | 4 |
| 2. | OBJE | ECTIVES | 4 |
| 2. | 1 | Primary Objective | 4 |
| | 2.2 | Secondary Objective | 4 |
| 3. | STUE | DY DESIGN | 5 |
| | 3.1 | Description of the Study | 5 |
| | 3.2 | Rationale for Study Design | 5 |
| | 3.3 | Outcome Measures | 5 |
| | | 3.3.1 Primary Outcome Measures | 5 |
| | | 3.3.2 Secondary Outcome Measures | 6 |
| | 3.4 | Safety Plan | 6 |
| | 3.5 | Compliance with Laws and Regulations | 7 |
| 4. | MATE | ERIALS AND METHODS | 7 |
| | 4.1 | Subjects | 7 |
| | | 4.1.1 Subject Selection | 7 |

## TABLE OF CONTENTS (cont'd)

| | | | | Fage |
|---|---|---|---|---|
| 4. | MATE | ERIALS A | AND METHODS (cont'd) | |
| | | 4.1.2 | Inclusion Criteria | 7 |
| | | 4.1.3 | Exclusion Criteria | 8 |
| | 42 | Method | of Treatment Assignment | 8 |
| | 4.3 | | Freatment | 9 |
| | | 4.3.1 | Formulation | 9 |
| | | 4.3.2 | Dosage, Administration, and Storage | 9 |
| | 4.4 | Concor | mitant and Excluded Therapies | 10 |
| | 4.5 | Study A | Assessments | 10 |
| | | 4.5.1 | Assessments during the Treatment Period | 10 |
| | | 4.5.2 | Early Termination Assessments | 11 |
| | 4.6 | Subject | t Discontinuation | 11 |
| | 4.7 | Study [ | Discontinuation | 12 |
| | 4.8 | Statistic | cal Methods | 12 |
| | | 4.8.1 | Analysis of the Conduct of the Study | 12 |
| | | 4.8.2 | Safety Analyses | 13 |
| | | 4.8.3 | Efficacy Analyses | 13 |
| | | 4.8.4 | Missing Data | 13 |
| | | 4.8.5 | Interim Analyses | 13 |
| | 4.9 | Data Q | uality Assurance | 14 |
| 50 | ASSE | SSMEN | T OF SAFETY | 14 |
| | 5.1 | Advers | e Events | 14 |
| | 5.2 | Baselin | e Medical Conditions | 15 |
| | 5.3 | Evaluat | tions | 15 |
| | 5.4 | Vital Si | gns | 16 |
| | 5.5 | Proced | ures for Recording and Reporting Adverse Events | 16 |
| | | 551 | Recording Adverse Events | 16 |
| | | 5.5.2 | Serious Adverse Events | 17 |
| | | 5.5.3 | Special Reporting Situations | 18 |
| | | 5.5.4 | Type and Duration of Follow-up After Adverse Events | 18 |
| | | 5.5.5 | Regulatory Reporting Requirements for Principal Investigator | rs |
| | | Holding | Their Own INDs | 19 |
| | | | 5.5.5.1 MedWatch 3500A Reporting Guidelines | 21 |

## TABLE OF CONTENTS (cont'd)

| | | | Page |
|---|---|---|---|
| 6. | INVES | STIGATOR REQUIREMENTS | 22 |
| | 6.1 | Study Initiation | 22 |
| | 6.2 | Study Completion | 23 |
| | 6.3 | Informed Consent Form | 23 |
| | 6.4 | Institutional Review Board or Ethics Committee Approval | 25 |
| | 6.5 | Case Report Forms. | 25 |
| | 6,6 | Study Drug Accountability | |
| | 6.7 | Disclosure of Data | |
| | 6.8 | Retention of Records | |
| REF | EREN | CES | 27 |
| APP | ENDIC | | |
| App | endix A | Study Flowchart | 28 |
| Арр | endix B | : Pre-Injection Procedures for All Subjects | 29 |
| Арре | endix C | : MedWatch Form FDA 3500A | 31 |
| Anne | endix D | Analysis of Similar Events | 33 |

## 1. BACKGROUND

## 1.1 PATHOPHYSIOLOGY

Diabetes is a disease of abnormal blood glucose secondary to insufficient or deficient insulin. This excess glucose is converted into alcohols through the aldose reductase pathway in tissues, the retina in particular because of the high level of aldose reductase in retinal capillaries. These alcohols result in structural changes in the capillaries that weaken them. This leads to microaneurysms, hemorrhages, increased permeability, and eventual closure of the capillaries. This results in hypoxia that causes several changes in the vasculature of the retina, including venous dilatation and new vessel growth. Areas of ischemic retina produce vasoproliferative substances, like vascular endothelial growth factor (VEGF). This stimulates the growth of new blood vessels in the retina, leading to neovascularization and proliferative diabetic retinopathy. (Aiello et al. 1999, Davis 1994)

## 1.2 TREATMENT OF DIABETIC NEOVASCULARIZATION

The current treatment of diabetic peripheral neovascularization is with panretinal photocoagulation. Laser photocoagulation is used to place 1200 or more 500-μm burns, separated by one-half burn width. Treatment is divided into two or more sessions. (ETDRS Report 9. 1991)

## 1.3 RANIBIZUMAB AND DIABETIC NEOVASCULARIZATION

Vascular endothelial growth factor A (VEGF-A) has been implicated in the development of neovascularization in diabetes. Using ranibizumab, an anti-VEGF-A drug, would inhibit this production.

## 1.4 NONCLINICAL EXPERIENCE WITH RANIBIZUMAB

## 1.4.1 Nonclinical Pharmacokinetics

The pharmacokinetics of ranibizumab have been investigated in rabbits and cynomolgus monkeys following intravitreal and intravenous administration. In

both species, following intravitreal administration, ranibizumab was cleared from the vitreous humor with a half-life of 2–3 days. Following single intravitreal administration to cynomolgus monkeys, retinal concentrations of ranibizumab were approximately one-third of vitreous concentrations and declined in parallel with vitreous concentrations. Intravitreal injections of ranibizumab can lead to detectable antibodies in serum in rabbits and cynomolgus monkeys.

## 1.4.2 Nonclinical Toxicology

A series of nonclinical studies of ranibizumab administered by intravitreal injection to cynomolgus monkeys have been performed (details regarding study design and results can be found in the Investigator Brochure).

## 1.4.3 Stability Studies

The stability of ranibizumab alone and in combination with verteporfin was assessed in vitro. The combination of ranibizumab and verteporfin in a 5% glucose solution at concentrations of 500 µg/mL and 1.4 µg/mL, respectively, resulted in ranibizumab degradation and a decrease in ranibizumab capacity to bind VEGF. The ranibizumab degradation products have not been fully characterized. Although it is currently unknown if such degradation also occurs in vivo, sequential administration of verteporfin followed by ranibizumab with an intervening washout period will decrease the likelihood of loss of ranibizumab activity and degradation.

## 1.5 CLINICAL EXPERIENCE WITH RANIBIZUMAB

Ranibizumab has been or is being clinically evaluated in eight wet AMD studies (additional details regarding study design and results can be found in the Investigator Brochure).

## 1.5.1 Study FVF1770g

The first clinical trial with ranibizumab, Study FVF1770g was a Phase Ia study of the molecule given as a single intravitreal injection to subjects with neovascular AMD. The goals of the study were to investigate safety and tolerability and to define the maximally tolerated dose (MTD). The single intravitreal MTD was determined to be 0.5 mg (limited by ocular inflammation).

## 1.5.2 Study FVF2128g

The Phase I/II study FVF2128g was the first clinical trial of multiple-dose regimens of intravitreally-administered ranibizumab. Sixty-four subjects were enrolled in the study. Data show that ranibizumab was safe and potentially efficacious in subjects with subfoveal choroidal neovascularization due to AMD.

## 1.5.3 Study FVF2425g

Study FVF2425g was a Phase I, open-label, randomized study of three escalating multiple-dose regimens of intravitreally-administered ranibizumab. Data show that doses of ranibizumab up to 2 mg could be safely given as part of an escalating dose regimen to subjects with subfoveal choroidal neovascularization due to AMD.

## 1,5.4 Study FVF2428g

Study FVF2428g is an ongoing Phase I/II, single-masked, multicenter study of the safety, tolerability, and efficacy of multiple-dose intravitreal injections of ranibizumab in combination with verteporfin PDT in subjects with neovascular AMD.

Preliminary findings from Study FVF2428g suggest that administration of ranibizumab injections 7 days ( $\pm 2$  days) after treatment with verteporfin PDT in the same eye may result in a decrease in visual acuity of  $\geq 30$  letters due to temporary intraocular inflammation (uveitis).

## 1.5.5 Study FVF2508g

Study FVF2508g is an ongoing Phase I extension study designed to assess the safety and tolerability of multiple-dose intravitreal injections of ranibizumab administered monthly in subjects who have completed the treatment phase of a Genentech-sponsored Phase I study.

## 1.5.6 Study FVF2587g

Study FVF2587g is an ongoing Phase III active treatment–controlled study designed to assess the efficacy and safety of intravitreal administered ranibizumab compared with verteporfin in subjects with angiographically determined, predominantly classic subfoveal neovascular AMD.

## 1.5.7 Study FVF2598g

Study FVF2598g is an ongoing Phase III study designed to assess the efficacy and safety of intravitreal injections of ranibizumab administered monthly compared with sham injections administered monthly in subjects with angiographically determined, minimally classic or occult subfoveal neovascular AMD.

## 1.5.8 Study FVF3192g

Study FVF3192g is an ongoing Phase IIIb study designed to assess the efficacy and safety of intravitreal injections of ranibizumab administered as three monthly injections followed by quarterly injections for a total duration of

24 months, in subjects with angiographically determined subfoveal neovascular AMD with or without classic CNV.

## 2. OBJECTIVES

## 2.1 Primary Objective

To compare the efficacy of ranibizumab versus additional panretinal photocoagulation on diabetic neovascularization that is persistent despite previous treatment with panretinal photocoagulation.

## 2.2 Secondary Objectives

To evaluate concomitant macular edema after intravitreal injection of ranibizumab in patients with persistent neovascularization.

## 3. STUDY DESIGN

## 3.1 DESCRIPTION OF THE STUDY

This is an open-label, Phase I/II study of intravitreally-administered ranibizumab in subjects with persistent (greater than three months) diabetic neovascularization previously treated with panretinal photocoagulation (at least 1200 or more 500-µm burns).

Consented, enrolled subjects will either receive open-label intravitreal injections of 0.5-mg dose of ranibizumab or additional panretinal photocoagulation (up to 500 300-500µm laser spots) in a ratio of two-to-one (2:1) at the beginning of the study period. ETDRS best-corrected visual acuity, contrast sensitivity, and Optos color photography will be performed at enrollment, at weeks 1, 2, 3 and 4, and at months 2, 3, 4, 5 and 6. The subjects will undergo fluorescein angiography utilizing the Optomap FA (fluorescein angiography) system and optical coherence tomography (OCT) at enrollment, at weeks 2 and 4, and at months 2, 3, 4 and 6. The subjects will be followed for a 6-month period for stabilization, regression, or recurrence of

neovascularization. In addition, patients will be evaluated for occurrence of macular edema.

### 3.2 RATIONALE FOR STUDY DESIGN

The pathophysiology of neovascularization associated with proliferative diabetic retinopathy has been shown to be via production of VEGF-A by ischemic retinal tissue. VEGF-A is produced and can be found in the vitreous cavity where it then acts to promote neovascularization. Ranibizumab is an anti-VEGF-A drug that has been shown to bind and inhibit the action of VEGF-A. Since diabetic neovascularization is the result of VEGF-A in the vitreous cavity, intravitreal injection of ranibizumab would bind the VEGF-A produced by the ischemic retina and therefore prevent neovascularization.

#### 3.3 OUTCOME MEASURES

## 3.3.1 Primary Outcome Measures

The primary efficacy outcome measures include:

- The percentage change of the area of the patient's neovascularization as measured in pixels by Optomap FA
- The percentage change of macular edema measured by retinal thickness by OCT

The primary safety and tolerability outcome measures are:

- Incidence and severity of ocular adverse events, as identified by ophthalmic examination
- Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs

## • 3.3.2 <u>Secondary Outcome Measures</u>

The secondary outcome measures are:

- Mean change in Best Corrected Visual Acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters 3 and 6 months
- Percentage of patients gaining 3 or more lines of vision according to
   ETDRS eye chart testing
- Occurrence rate of proliferative diabetic complications including vitreous hemorrhage, iris neovascularization and tractional retinal detachment

#### 3.4 SAFETY PLAN

The safety assessments to be conducted for this study are listed in Section 4.5 and Appendix A.

- Potential adverse events include but are not limited to local injection site reaction, subconjunctival hemorrhage, vitreous hemorrhage, retinal tear or detachment or endophthalmitis.
- If a patient has an occurrence of retinal tear or detachment or endophthalmitis:
  - The patient will not be included in the study
  - Treatment will be based on the event and at the discretion of the treating physician based on current accepted practice standards
  - Any necessary testing such as ultrasound or cultures will be performed as indicated by the specific event.
  - Any necessary procedures, such as vitreous tap and injection,
     laser for tears or surgical repair of detachments will be performed
     according to current practice standards

## 3.5 COMPLIANCE WITH LAWS AND REGULATIONS

This study will be conducted in accordance with current U.S. Food and Drug Administration (FDA) Good Clinical Practices (GCPs), and local ethical and legal requirements.

## 4. MATERIALS AND METHODS

#### 4.1 SUBJECTS

## 4.1.1 Subject Selection

Ten (10) subjects from one site in the United States will be enrolled. Eligible subjects will have provided informed consent. (See Appendix A, the study flow chart, for screening assessments.)

## 4.1.2 Inclusion Criteria

Subjects will be eligible if the following criteria are met:

- Ability to provide written informed consent and comply with study assessments for the full duration of the study
- Age ≥ 18 years
- Patient-related considerations

Patients with Diabetes Mellitus (Type I or II) are eligible. HgA<sub>1c</sub> will be evaluated at the beginning of the study, but this value will have no significance in inclusion or exclusion. Patients will not be pregnant at enrollment and must provide evidence of the use of two types of birth control while enrolled in the study. Patients will have no known sensitivity to ranibizumab or other anti-VEGF injections.

## Disease-related considerations

Patients will have diabetic neovascularization as seen on fluorescein angiography that was previously treated with full (at least 1200 laser burns) panretinal photocoagulation and that has persisted at least three months. There will be no evidence of ocular inflammation at enrollment. There is no restriction on patient's current medications or concomitant illnesses as long as there is no interference with patient follow-up.

#### Other considerations

Patients may not be enrolled in another clinical study or observational trial. There is no limitation on patient's institutional status as long as the patient is able to participate in follow-up.

## 4.1.3 Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

- Pregnancy (positive pregnancy test)
- Uncontrolled glaucoma on three medicines or more to control intraocular pressure
- Prior enrollment in the study
- Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
- Participation in another simultaneous medical investigation or trial

## 4.2 METHOD OF TREATMENT ASSIGNMENT

The enrolled subjects will be randomized into two groups, 0.5 mg injection of ranibizumab or additional panretinal photocoagulation (PRP), in a two-to-one ratio (2:1). Randomization will occur by alternating treatment groups in the above ratio, as patients are included in the study. For example, Patient A and

Patient B will receive ranibizumab, Patient C will receive additional PRP,
Patient D and Patient E will receive ranibizumab, etc. Therefore, seven (7)
patients will receive ranibizumab and three (3) patients will receive additional
PRP. There will be no masking of which treatment each patient receives.

#### 4.3 STUDY TREATMENT

## • 4.3.1 Formulation

Ranibizumab is formulated as a sterile solution aseptically filled in a sterile, 3-mL stoppered glass vial. Each vial contains 0.5 mL of 10mg/mL (0.5-mg dose level) ranibizumab aqueous solution (pH 5.5) with histidine, trehalose, and polysorbate 20. The vial contains no preservative and is suitable for single use only.

For further details and molecule characterization, see the Investigator Brochure.

## 4.3.2 Dosage, Administration, and Storage

#### a. Dosage

0.5-mg of ranibizumab will be injected intravitreally at the patient's enrollment in the study for patients in the ranibizumab treatment group.

## b. Administration

\*See Appendix B for detailed pre-injection procedures.

## c. Storage

Upon receipt, study drug kits should be refrigerated at 2°C - 8°C (36°F - 46°F). DO NOT FREEZE. Do not use beyond the expiration date. Ranibizumab vials should remain refrigerated. Protect vials from direct sunlight.

VIALS ARE FOR SINGLE USE ONLY. Vials used for one subject may not be used for any other subject.

## 4.4 CONCOMITANT AND EXCLUDED THERAPIES

Subjects may continue to receive all medications and standard treatments administered for their conditions at the discretion of their treating physician.

## 4.5 STUDY ASSESSMENTS

## 4.5.1 Assessments during the Treatment Period

## **Enrollment**

- Informed consent
- Demographic data
- Hemoglobin A1c
- Urine pregnancy test
- Physical examination and medical history
- Vital signs
- Intraocular pressure
- Slit-lamp exam
- Dilated binocular indirect ophthalmoscopy
- Ranibizumab treatment with finger count vision after injection OR Panretinal photocoagulation (up to 500 300-500μm laser spots)
- Telephone safety check (2 days after visit)
- SAE monitoring
- ETDRS BCVA at 4 meters
- Contrast sensitivity testing
- Optomap FA
- Optical Coherence Tomography
- Optos color photos

## 1 week, 3 weeks, and 5 months

Vital signs

Protocol: FVF3817s Final

11

- Intraocular pressure
- Slit-lamp exam
- Dilated binocular indirect ophthalmoscopy
- SAE monitoring
- ETDRS BCVA at 4 meters
- · Contrast sensitivity testing
- Optos color photos

## 2 and 4 weeks, 2, 3, 4 and 6 months

- Vital signs
- Intraocular pressure
- Slit-lamp exam
- Dilated binocular indirect ophthalmoscopy
- SAE monitoring
- ETDRS BCVA at 4 meters
- · Contrast sensitivity testing
- Optomap FA
- Optical Coherence Tomography
- Optos color photos

## 4.5.2 Early Termination Assessments

Subjects who withdraw from the study prior to completion should return for an early termination evaluation 14 days (± 7 days) following the last injection/study visit for monitoring of all adverse events (serious and nonserious). The schedule of assessments for early termination is the same as that for the final visit.

#### 4.6 SUBJECT DISCONTINUATION

Subjects have a right to withdraw from the study at any time.

The subject may be withdrawn from the study for any reasons: if it is in the best interest of the subject, intercurrent illness, adverse events, or worsening

Protocol: FVF3817s Final

12 28DEC06

condition. Rush University Medical Center may request the withdrawal of a subject because of protocol violations, administrative reasons, or any other valid and ethical reasons.

Subjects will be discontinued and receive standard additional panretinal photocoagulation for development of neovascular glaucoma (NVG).

Other reasons for subject discontinuation may include, but are not limited to, the following:

- Sensory rhegmatogenous retinal detachment or Stage 3 or 4 macular hole
- Investigator determination that it is not in the best interest of the subject to continue participation
- Pregnancy
- Verteporfin PDT treatment in the study eye
- Pegaptanib sodium injection treatment in either eye
- SAE
- Any other safety concerns

If a subject discontinues or is discontinued from the study, he or she will not be allowed to re-enter the study.

In the event of an adverse event in the study eye that is considered by the investigator to be severe in intensity, serious consideration should be given to discontinuing the subject from the study.

#### 4.7 STUDY DISCONTINUATION

This study may be terminated by Rush University Medical Center at any time. Reasons for terminating the study may include the following:

- The incidence or severity of adverse events in this or other studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Data recording is inaccurate or incomplete

#### 4.8 STATISTICAL METHODS

## 4.8.1 Analysis of the Conduct of the Study

There is no formal sample size calculation in this pilot study. As this is a phase I/II study, a sample size of 10 patients is chosen, making sure that it is feasible financially to conduct the study and logistically to complete the study within 12 months. If and when the study is planned for a phase II randomized control trial, appropriate statistical analysis will be determined.

## • 4.8.2 Safety Analyses

Any adverse events, laboratory assessments, physical examinations, vital signs, ocular examinations and measurements from all 10 subjects will be utilized to summarize safety data for this pilot study.

## 4.8.3 <u>Efficacy Analyses</u>

As this is a small pilot study, no formal statistical analyses are planned

## a. Primary Endpoint

- The percentage change of the area measured in pixels of the patient's neovascularization as measured by Optomap FA fluorescein angiography
- The percentage change of macular edema measured by retinal thickness by OCT

## b. Secondary Endpoints

 Mean change in Best Corrected Visual Acuity (BCVA), as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 4 meters, at 3 and 6 months  Percentage of patients gaining 3 or more lines of vision according to ETDRS eye chart testing

 Occurrence rate of proliferative diabetic complications including vitreous hemorrhage, iris neovascularization and tractional retinal detachment

## 4.8.4 Missing Data

Analyses of efficacy and safety will be based on available cases, without imputation for missing values.

## 4.8.5 Interim Analyses

No formal schedule of interim analyses is planned. Reports of adverse events from this extension study may be reviewed and summarized periodically while the study is ongoing to ensure the safety of subjects.

#### 4.9 DATA QUALITY ASSURANCE

Accurate, consistent, and reliable data will be ensured through the use of standard practices and procedures.

## 5. ASSESSMENT OF SAFETY

The safety of ranibizumab will be assessed through the collection and analysis of any adverse events that occur during the study whether related to the study drug or not.

#### 5.1 ADVERSE EVENTS

AEs that start on Day 0 through the last study visit will be recorded on the appropriate AE pages of the CRF. Subjects discontinuing early from the study should return for an early termination evaluation and will be contacted 7 days after their last injection or study visit to elicit for occurrence of adverse events (serious and nonserious).

For this protocol, an AE is any "on study" untoward medical occurrence (e.g., sign, symptom, disease, syndrome, intercurrent illness) that occurs in a study subject, regardless of the suspected cause. "On study" refers to Day 0 through the last study visit.

Unchanged, chronic conditions are NOT AEs and should not be recorded on the AE pages of the CRF. An exacerbation or worsening of a chronic condition should be recorded as an AE.

Both serious and nonserious AEs should be graded on a three-point scale (mild, moderate, severe) and reported in detail on the appropriate AE page of the CRF.

The suggested definitions are as follows:

Mild: Discomfort noticed but no disruption of normal daily activity

Moderate: Discomfort sufficient to reduce or affect normal daily activity

Severe: Incapacitating with inability to work or perform normal daily activity

Using the following criteria, investigators also need to assess whether there is a reasonable possibility that study drug caused or contributed to the AE.

Yes (possibly or probably)

There is a clinically plausible time sequence between onset of the AE and study drug administration; and/or

There is a biologically plausible mechanism for study drug causing or contributing to the AE; and

The AE may or may not be attributed to concurrent/underlying illness, other drugs, or procedures.

Protocol: FVF3817s Final

28DEC06

No.

A clinically plausible temporal sequence is inconsistent with the onset of the AE and study drug administration; and/or

A causal relationship is considered biologically implausible.

#### 5.2 BASELINE MEDICAL CONDITIONS

It is not necessary to complete an AE CRF page for chronic medical conditions present at enrollment that do not worsen in intensity or frequency during the trial. These medical conditions should be adequately documented on the appropriate page of the CRF (medical history and/or physical examination). However, medical conditions present at enrollment that worsen in intensity or frequency during the treatment or post-treatment periods and ongoing AEs that started during the previous study should be reported and recorded as AEs.

#### 5.3 EVALUATIONS

Reviews of body systems will be performed.

Ophthalmologic evaluations will include slit lamp examination, dilated binocular indirect high-magnification ophthalmoscopy, measurements of BCVA and intraocular pressure, and finger-count testing. (See Section 4.5 for a detailed description of the study assessments.)

#### 5.4 VITAL SIGNS

Pulse, blood pressure, respiration, and temperature will be measured at protocol-specified study visits (see Section 4.5).

## 5.5 PROCEDURES FOR RECORDING AND REPORTING ADVERSE EVENTS

## 5.5.1 Recording Adverse Events (see examples below)

To improve the quality and precision of acquired AE data, investigators should observe the following guidelines:

- Whenever possible, use recognized medical terms when recording AEs on the AE pages of the CRF. Do not use colloquialisms and/or abbreviations.
- If known, record the diagnosis (i.e., disease or syndrome) rather than
  component signs and symptoms on AE pages of the CRF (e.g., record
  congestive heart failure rather than dyspnea, rales, and cyanosis).
  However, signs and symptoms that are considered unrelated to an
  encountered syndrome or disease should be recorded as individual AEs
  on the CRF (e.g., if congestive heart failure and severe headache are
  observed at the same time, each events should be recorded as an
  individual AE).
- AEs occurring secondary to other events (e.g., sequelae) should be identified by the primary cause. A "primary" AE, if clearly identifiable, generally represents the most accurate clinical term to record on AE pages of the CRF. If a primary serious AE (SAE) is recorded on an SAE CRF, events occurring secondary to the primary event should be described in the narrative description of the case.

For example:

Orthostatic hypotension

→ Fainting and fall to floor

→ Head trauma → Neck pain

The primary AE is orthostatic hypotension.

## 5.5.2 Serious Adverse Events

An AE occurring **at any dose** (including overdose) should be classified as **SERIOUS** if:

- It resulted in death (i.e., the AE caused or led to death).
- It was life threatening (i.e., the AE placed the subject at immediate risk
  of death; it does not apply to an AE that hypothetically might have
  caused death if it were more severe).
- It required or prolonged inpatient hospitalization (i.e., the AE required at least a 24-hour inpatient hospitalization or prolonged a hospitalization beyond the expected length of stay; hospitalizations for elective medical/surgical procedures, scheduled treatments, or routine checkups are not SAEs by this criterion).
- It was disabling (i.e., the AE resulted in a substantial disruption of the subject's ability to carry out normal life functions).
- It resulted in a congenital anomaly/birth defect (i.e., an adverse
  outcome in a child or fetus of a subject exposed to the molecule or
  study drug prior to conception or during pregnancy).
- It does not meet any of the above serious criteria but may jeopardize
  the subject or may require medical or surgical intervention to prevent
  one of the outcomes listed above.

## **SAE Reporting**

Investigators must report all SAEs to Genentech within 48 hours of observing or learning of the event. For initial SAE reports, investigators should record all case details that can be gathered within 48 hours on the SAE page of the CRF.

The completed SAE page and SAE Fax Cover Sheet should be faxed immediately upon completion to the Genentech Drug Safety at:

(650) 225-4682

or

(650) 225-5288

Relevant follow-up information should be submitted to Genentech as soon as it becomes available.

## 5.5.3 <u>Special Reporting Situations</u>

#### a. Death

Death is an outcome of an event. The **event** that resulted in the death should be recorded and reported on the SAE pages of the CRF.

## b. Hospitalizations for Surgical or Diagnostic Procedures

The **illness** leading to the surgical or diagnostic procedure should be recorded as the SAE, not the procedure itself. The procedure should be captured in the case narrative as part of the action taken in response to the illness.

## c. Pregnancy

## 5.5.4 Type And Duration Of Follow-Up After Adverse Events

All reported AEs should be followed until resolution or until the subject's participation in the study ends. Subjects who have an ongoing study drug—related SAE at study completion or at discontinuation from the study will be followed by the investigator or his or her designee until the event is resolved or determined to be irreversible, chronic, or stable by the investigator.

# • <u>5.5.5 Regulatory Reporting Requirements for Principal Investigators Holding</u> Their Own INDs

Investigators conducting studies under their own INDs are responsible for expedited Safety Reports and IND Annual Reports to the FDA.

## **Expedited IND Safety Reports:**

For this **Investigator Sponsored IND Study**, some additional reporting requirements for the FDA apply in accordance with the guidance set forth in 21 CFR § 312.32.

Events meeting the following criteria should be submitted to the Food and Drug Administration (FDA) as expedited IND Safety Reports according to the following guidance and timelines:

## Fatal or Life-Threatening, Unexpected, Drug-related SAEs

The Investigator is required to notify the FDA of any <u>fatal or life-threatening</u> adverse event that is <u>unexpected</u> and assessed by the investigator to be <u>related</u> to the use of ranibizumab. Reports are to be telephoned or faxed to the FDA <u>within 7 calendar days</u> of the Investigator's knowledge of the event. Additionally, notify Genentech Medical Science Liaison by telephone <u>within 7</u> calendar days.

An <u>unexpected</u> adverse event is one that is not already described in the ranibizumab Investigator's Brochure (IB) This includes adverse events that have not been identified as life-threatening or causing a death as described in the IB, for example, elevated hepatic enzymes or hepatitis versus liver failure. This also includes unusual AEs not specifically described in the IB, for example, hemorrhage versus intraocular bleeding.

The 7-day telephone or fax report must be followed within 8 additional calendar days by a written IND safety report (MedWatch 3500A Form). Written IND Safety Reports should include an Analysis of Similar Events in accordance with regulation 21 CFR § 312.32. (See Appendix D for Analysis of Similar Events template). All safety reports previously filed to the IND concerning similar events should be analyzed. The significance of the new report in light of the previous, similar reports should be commented on.

Written IND safety reports with Analysis of Similar Events are to be submitted to the FDA, Genentech, the IRB, and all participating investigators within 15 calendar days of the

Investigator's knowledge of the event. The FDA prefers these reports on a MedWatch 3500A Form but alternative formats are acceptable (e.g. summary letter).

## FDA Fax Number for IND Safety Reports:

1 (800) 332-0178

## All written IND Safety Reports submitted to the FDA by the Investigator must also be faxed to:

Genentech Medical Science Liaison:

Name: Sara L. Butterworth, OD, FAAO Tel: (319) 358-9770 or (319) 331-9795)

Fax: (319) 354-4751

#### AND:

Genentech Drug Safety at:

(650) 225-4682 or (650) 225-5288

#### AND:

Institutional Review Board:

Research and Clinical Trials Administration Office Rush University Medical Center 1725 W. Harrison, Suite 439 Chicago, IL 60612 Phone: (312) 942-5498

Fax: (312) 942-2874

For questions related to Safety reporting, contact your Genentech Medical Science Liaison.

## Serious, Unexpected, and Drug-related SAEs (not life-threatening or fatal)

A written IND Safety Report (described above) should also be produced for any unexpected SAE that is considered <u>related</u> to the use of ranibizumab but is <u>not life-threatening or fatal</u>. Investigators are required to notify the FDA, Genentech, the IRB, and all participating investigators by submitting the IND Safety Report within 15 days of the Investigator's knowledge of the event.

Protocol: FVF3817s Final

28DEC06

**IND Annual Reports** 

All IND annual reports submitted to the FDA by the Investigator should be copied to Genentech. Copies of such reports should be mailed to:

Jim Nickas
Director of Drug Safety
Mailstop #84
Genentech, Inc.
1 DNA Way
South San Francisco, CA 94080-4990

# <u>5.5.5.1 MedWatch 3500A Reporting Guidelines: (See Appendix C for MedWatch form)</u>

In addition to completing appropriate patient demographic and suspect medication information, the report should include the following information within the Event Description (section 5) of the MedWatch 3500A form:

- Identification of the primary event term
- Protocol description (and number, if assigned)
- Description of event, severity, treatment, and outcome if known
- Supportive laboratory results and diagnostics
- Investigator's assessment of the relationship of the adverse event to each investigational product and suspect medication
- If a death occurred, autopsy results if available

MedWatch forms can be obtained on-line at <a href="www.fda.gov/medwatch">www.fda.gov/medwatch</a> or by calling the FDA at 1-800-332-1088.

## Follow-up information:

Additional information may be added to a previously submitted report by any of the following methods:

- Add to the original MedWatch 3500A report and submit it as follow-up
- Add documents and submit as follow-up with the original MedWatch 3500A form
- Summarize new information and fax it with a cover letter including subject identifiers (i.e. D.O.B. initial, subject number), protocol description and number, if assigned, brief adverse event description, and notation that additional or follow-up information is being submitted. (Patient identifiers are important so that new information is added to the correct initial report.)

Protocol: FVF3817s Final

28DEC06

Occasionally Genentech may contact the investigator for additional information, clarification, or current status of the subject for whom an adverse event was reported.

For questions regarding SAE reporting, you may contact the Genentech Medical Science Liaison.

## 6.0 INVESTIGATOR REQUIREMENTS

#### 6.1 STUDY INITIATION

Before the start of this study, the following documents must be on file with Rush University Medical Center or its appointed representative:

- FDA correspondence letter assigning an IND number or an IND waiver letter
- Original U.S. FDA Form 1572 (for all studies conducted under U.S. Investigational New Drug [IND] regulations), signed by the Principal Investigator
- The names of any sub-investigators must appear on this form.
   Investigators must also complete all regulatory documentation as required by local and national regulations.
- Current curricula vitae of the Principal Investigator
- Written documentation of IRB approval of protocol (identified by Rush University Medical Center, protocol number or title and date of approval) and informed consent document (identified by Rush University Medical Center protocol number or title and date of approval)
- A copy of the IRB-approved informed consent document
- Written documentation of IRB review and approval of any advertising materials to be used for study recruitment, if applicable
- The informed consent document and any advertising materials must also be reviewed and approved by the Rush University Medical Center Legal Department.

- Certified translations of IRB approval letters, pertinent correspondence, and approved informed consent document (when applicable)
- Current laboratory certification of the laboratory performing the analysis as well as current normal laboratory ranges for all laboratory tests.

#### 6.2 STUDY COMPLETION

The following data and materials are required by Rush University Medical Center before a study can be considered complete or terminated:

- Laboratory findings, clinical data, and all special test results from screening through the end of the study follow-up period (if applicable)
- Case Report Forms properly completed by appropriate study personnel and signed and dated by the investigator (if applicable)
- Copies of protocol amendments and IRB approval/notification (if applicable)
- A summary of the study prepared by the Principal Investigator (will accept IRB summary close letter) (if applicable)
- All regulatory documents (e.g., curricula vitae for each Principal Investigator, U.S. FDA Form 1572)

#### 6.3 INFORMED CONSENT

Informed consent documents will be provided to each subject.

The informed consent document must be signed and dated by the subject or the subject's legally authorized representative before his or her participation in the study. The case history for each subject shall document that informed consent was obtained prior to participation in the study. A copy of the informed consent document must be provided to the subject or the subject's legally authorized representative. If applicable, it will be provided in a certified translation of the local language.

Protocol: FVF3817s Final

25 28DEC06

Signed consent forms must remain in each subject's study file and must be available for verification at any time.

The following basic elements must be included:

- A statement that the study involves research, an explanation of the purposes of the research and the expected duration of the patient's participation, a description of the procedures to be followed, and identification of any procedures or drug used for purposes which are experimental
- A description of any reasonably foreseeable risks or discomforts to the patients
- A description of any benefits to the patient or to others which may reasonably be expected from the research. A description that there may be no benefit from this research.
- A disclosure of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the patient
- A statement describing the extent, if any, to which confidentiality records identifying the patient will be maintained and that notes the possibility that the FDA and Rush University Medical Center and the drug manufacturer may inspect the records
- For research involving more than minimal risk, an explanation as to whether any compensation and any medical treatments are available should injury occur and, if so, what they consist of or where further information may be obtained
- An explanation of whom to contact for answers to pertinent questions about the research and research patient's rights, and whom to contact in the event of a research-related injury to the patient
- A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the patient is otherwise entitled, and that the patient may discontinue participation at any time

without penalty or loss of benefits to which the patient is otherwise entitled

## 6.4 INSTITUTIONAL REVIEW BOARD OR ETHICS COMMITTEE APPROVAL

This protocol, the informed consent document, and relevant supporting information must be submitted to the IRB/EC for review and must be approved before the study is initiated. The study will be conducted in accordance with U.S. FDA, applicable national and local health authorities, and IRB/EC requirements.

The Principal Investigator is responsible for keeping the IRB/EC apprised of the progress of the study and of any changes made to the protocol as deemed appropriate, but in any case the IRB/EC must be updated at least once a year. The Principal Investigator must also keep the IRB/EC informed of any significant adverse events.

Investigators are required to promptly notify their respective IRB/EC of all adverse drug reactions that are both serious and unexpected. This generally refers to serious adverse events that are not already identified in the Investigator Brochure and that are considered possibly or probably related to the study drug by the investigator. Some IRBs or ECs may have other specific adverse event requirements that investigators are expected to adhere to Investigators must immediately forward to their IRB/EC any written safety report or update provided by Rush University Medical Center (e.g., IND safety report, Investigator Brochure, safety amendments and updates, etc.).

#### 6.5 CASE REPORT FORMS

All CRFs should be filled out completely by appropriate personnel. The CRF should be reviewed, signed, and dated by the investigator.

All CRFs should be completed in a neat, legible manner to ensure accurate interpretation of data. Black ink is required to ensure clarity of reproduced CRF copies. When making changes or corrections, cross out the original entry with a single line, and initial and date the change. DO NOT ERASE, OVERWRITE, OR USE CORRECTION FLUID ON THE ORIGINAL.

#### 6.6 STUDY DRUG ACCOUNTABILITY

The Investigator is responsible for the control and distribution of study drug.

All partially used or empty containers should be disposed of at the study site according to institutional standard operating procedure.

## 6.7 DISCLOSURE OF DATA

Subject medical information obtained by this study is confidential, and disclosure to third parties other than those noted below is prohibited.

Upon the subject's permission, medical information may be given to his or her personal physician or other appropriate medical personnel responsible for his or her welfare.

Data generated by this study must be available for inspection upon request by representatives of the U.S. FDA, national and local health authorities, the drug manufacturer and the IRB/EC for each study site, if appropriate.

## 6.8 RETENTION OF RECORDS

U.S. FDA regulations (21 CFR §312.62[c]) require that records and documents pertaining to the conduct of this study and the distribution of investigational drug, including CRFs, consent forms, laboratory test results, and medication inventory records, must be retained by the Principal Investigator for 2 years after the investigation is discontinued and the U.S. FDA and the applicable national and local health authorities are notified.

#### **REFERENCES**

Aiello LM, Cavallerano JD, Aiello LP, Bursell SE: Diabetic retinopathy. In: Guyer DR, Yannuzzi LA, Chang S, Shields JA, Green WR, eds. Retina Vitreous Macula. Vol 2. 1999:316-344.

Davis MD: Proliferative diabetic retinopathy. In: Ryan SJ, ed. Retina. Vol 2. 1994:1319-1360

Early photocoagulation for diabetic retinopathy. ETDRS report 9. Early Treatment

Diabetic Retinopathy Study Research Group. Ophthalmology. 1991;98: 766-785

Protocol: FVF3817s Final

29 28DEC06

| | Enrollment | 1 week | 2 weeks | 3 weeks | 4 weeks | 2 months | 3 months | 4months | 5 months | 6 months | 14 Days after<br>withdrawal |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Intormed consent | × | | | | | | | | | | |
| Demographic data | × | | | | | | | | | | |
| Hemoglobin A <sub>1C</sub> | × | | | | | | | | | | |
| Urine Pregnancy Test | × | | | | | | | | | | |
| Physical examination and medical history | × | | | | | | | | | | |
| Vital signs | × | × | × | × | × | × | × | × | × | × | × |
| Infraocular Pressure | × | × | × | × | × | × | × | × | × | × | × |
| Slit-lamp exam | × | × | × | × | × | × | × | × | × | × | × |
| Dilated binocular indirect ophthalmoscopy | × | × | × | × | × | × | × | × | × | × | × |
| Ranibizumab treatment | ** | | | | | | | | | | |
| Finger count vision after injection | × | | | | | | | | | | |
| Panretinal photocoagulation | *X | | | | | | | | | | |
| Telephone Safety<br>Check | X+2Days | , | - | | | | | | | | |
| SAE monitoring | × | × | × | × | × | × | × | × | × | × | × |
| ETDRS BCVA at 4<br>meters | X | × | × | × | × | × | × | × | × | × | × |
| Contrast sensitivity testing | × | × | × | × | × | × | × | × | × | × | × |
| Optomap FA | × | | × | | × | × | × | × | | × | × |
| Optical Coherence<br>Tomography | × | | × | | × | × | × | × | | × | × |
| Optos color photos | × | × | × | × | × | × | × | × | × | × | × |
| * Patients will be treated with either ranibizumab or PRP_depending upon randomization | eated with eithe | r ranibizum | ah or PRP, de | pending upo | n randomiza | fion | | | | | |

<sup>\*</sup> Patients will be treated with either ranibizumab or PRP, depending upon randomization

#### APPENDIX B

## Pre-Injection Procedures for All Subjects

The following procedures will be implemented to minimize the risk of potential adverse events associated with serial intravitreal injections (e.g., endophthalmitis). Aseptic technique will be observed by clinic staff involved in the injection tray assembly, anesthetic preparation, and study drug preparation and administration. In addition to the procedures outlined below, added safety measures in adherence to specific institutional policies associated with intravitreal injections will be observed.

The following procedures (except where noted) will be conducted by the investigator. Subjects will have received antimicrobials (e.g. trimethoprim-polymyxin B ophthalmic solution, ofloxacin ophthalmic solution, ophthalmic gatifloxacin solution, ophthalmic moxifloxacin solution) for self-administration four times daily for 3 days prior to treatment.

- The technician assembles the supplies and prepares a sterile field. Supplies include 10% povidone iodine swabs, sterile surgical gloves, 4×4 sterile pads, pack of sterile cotton-tipped applicators, eyelid speculum, sterile ophthalmic drape, 0.5% proparacaine hydrochloride, 5% povidone iodine ophthalmic solution, 1% lidocaine for injection, ophthalmic antimicrobial solution (e.g. trimethoprim-polymyxin B ophthalmic solution, ofloxacin ophthalmic solution, ophthalmic gatifloxacin solution, ophthalmic moxifloxacin solution), and injection supplies.
- Instill 2 drops of 0.5% proparacaine hydrochloride into the study eye, followed by 2 drops of a broad-spectrum antimicrobial solution (e.g. trimethoprim-polymyxin B ophthalmic solution, ofloxacin ophthalmic solution, ophthalmic gatifloxacin solution, ophthalmic moxifloxacin solution).
- Disinfect the periocular skin and eyelid of the study eye in preparation for injection. Scrub the eyelid, lashes, and periorbital skin with 10% povidone iodine swabs, starting with the eyelid and lashes and continuing with the surrounding periocular skin. Make certain that the eyelid margins and lashes are swabbed, and proceed in a systematic fashion, from medial to temporal aspects.
- The investigator will glove, place sterile ophthalmic drape to isolate the field, and place the speculum underneath the eyelid of the study eye.
- Instill 2 drops of 5% povidone iodine ophthalmic solution in the study eye, making sure the drops cover the planned injection site on the conjunctiva.
- Wait 90 seconds.

- Saturate a sterile cotton-tipped applicator with 0.5% proparacaine hydrochloride drops and hold the swab against the planned intravitreal injection site for 10 seconds in preparation for the subconjunctival injection of 1% lidocaine hydrochloride ophthalmic solution for injection (without epinephrine).
- Use a sterile 4×4 pad in a single wipe to absorb excess liquid and to dry the periocular skin.

## APPENDIX C: MedWatch Form FDA 3500A

| The FDA Safety Information and | For use by us<br>importers, distributor | ser-facilities. | Mir Report≠ | | ı |
|---|---|---|---|---|---|
| The FDA Safety Information and | impostore distributor | | | | |
| | for MANDATS | es and manufacturers<br>ORY reporting | UF/Importer Rep | :crt# | |
| | Page | of | | | and they flack |
| Adverse Event Reporting Program | | C. SUSPECT MEDIC | ATTOMISS | | FDA ties Cob |
| A PATIENT INFORMATION | , sex 4. Weignt | 1. Name (Give (apeled siteria | | Orasikeř | |
| 5. Patlant Identifier 2. Age at Tame 5. of Event: | 4. 4121Qsib | 21 | | | |
| ar | Famaleips | ** | | | · |
| Defe<br>in confidence of Birth: | ∏ 2/siekgs | \$3 | | | aise (if unanown, give duration) |
| B. ADVERSE EVENT OR PRODUCT PROBLEM | | 2. Dogs, Frequency & Roule | i Çeed | | best estimate) |
| 5. Adverse Event under Froduct Problem (d.g., | | <b>#1</b> | | <b>‡1</b> | |
| | - Trickly-indubitations | #2 | | #2 | |
| Outdomes Attributed to Adverse Event Disability (Check of that apply) Occeptable | THE MANY IN | 4. Diagnosis for Use (Indias | ton) | | ivent Abaled After Use<br>Hopped or Dose Reduced? |
| i Centa: | ervandan to Prevent | <b>#1</b> | | - 1 | Mys Myn Do±snt |
| | moalment/Damag# | <b>#2</b> | | | Apply |
| Hospitalization - Initial or prolonged Chiner | | S. Loi# (Fension) | Exp. Date 68 kg | rown) #2 | Yes Mo Apply |
| | eport (movissy/year) | #1 | ±1 | | vent Reappeared After |
| S. Wall by Land (Managayers) | ., | #3 | #2 | | Reinfraduction? |
| 5. Decaribe Event of Problem | | 9. KDC# (For product probler | | | Appy |
| | | - | _ | <b>#</b> 2 | Yes No Desart |
| | | 13. Concemilant Medical Pr | ndustic and There | any Dates (Ex: | clude treatment of event) |
| | | D. SUSPECT MEDIC. 1. Stand Rame 2. Type of Device | AL DEVICE | | |
| | | - 1,2- | | | |
| | | 3. Manufasturer Name, Olly | and State | | |
| | | 4. Nacel # | £st≢ | | 5. Operator of Caylor Health Professions |
| | Printed and the second | Catalog # | | Date (mo/day | Lay User/Pallent |
| *** | | Serial # | Others | | |
| E. Rejevant TaccolLaboratory Dafa, including Sates | | 5. if implanted, Give Date in | | | d, Give Dale (ms/day)y() |
| | | 8. is into a Single-use Devic | e that was Repro | ecesed and R | egged on a Patient? |
| | | Yes No | Wame and Adde | ess of Bearon | 95501 |
| | | - 1 that the man late of Soley | | | |
| | | 13. Device Available for Eva | luation7 (Do not<br>Returned to Ma | | |
| | | 11. Concomitant Wedical Pro | | | anticativity |
| 7. Other Relevant Mictory, Including Proexisting Medical Condi-<br>race, cregnancy, smoking and alcohol use, nepaltorenal dysfun. | Ikiona (e.g. allergies,<br>Icitan. etc.) | 11. Соверным мевем на | 50854 <b>6-9</b> 26 (52) | apy Dates (23: | CHEC Properties of Laboration |
| | | | <b></b> | 11 (N. 17 A | g Sid Hoper Conference |
| | | E INDIAL REPORTE 1. Same and Address | Phone t | 1 | |
| | | <u>.</u> | <u> </u> | | |
| Code instance of a new of few | ant constitute | | | | |
| Submission of a report does an admission that medical product caused or contributed FORM FDA 3500A (9/03) | ersonnel, user<br>nanufacturer or | 2. Health Professional? 3. | Copupation | | 4. Indial Reporter Also Sens<br>Report to FDA Yes No Unk. |

Protocol: FVF3817s Final

33

28DEC06

## Medication and Device Experience Report

Submission of a report does not constitute an admission that medical personnel, user facility, importer, distributor, manufacturer or product caused or contributed to the event

U.S. DEPARTMENT OF HEALTH AND HUMAN SERVICES
PUBLIC HEALTH SERVICE - FOOD and Drug Administration
FILM USE OWLY

| (Consider) | | |
|---|---|---|
| Refer to guidelines for specific instructions. Page | | A COLUMN TO THE PARTY OF THE PA |
| F. FOR USE BY USER FACILITY/IMPORTER (Devices Only) | H, DEVICE MANUFACTURERS ONLY | |
| %. Check One Z. UFAmporlar Report Number | 1. Type of Reportable Event | 2. If Follow-up, What Type? |
| User Facility Impaner | S#SIN | ☐ Conesiøn |
| 2. User Facility or Importer Name/Address | Serious Wury | Adeilional information |
| | Malfurgion | Response is FDA Request |
| | Officer: | Device Exaligation |
| | | 4. Device Manufacture Date (mc//r) |
| | 3. Device Evaluated by Manutacturer? | 4. Daylor satisfication of process |
| | Not Renamed to Manufacturer | 1 |
| 4. Cardact Person 5. Phone Number | Yes Svehation Summary Atlached | €. Labeled for \$ingle Use? |
| | Wo (Attack page to explain why sel) at gravite code: | |
| 6. Date User Facility of 7. Type of Report 8. Date of Title Report (modds/f/f) | F121 22 222 | ☐ Yes ☐ N⊅ |
| Aware of Event (mostay/91) [ initial | | |
| = 50kg/m=x3 # | 5. Evaluation Ondes (Refer to coding manual) | |
| 5: Approximate 13. Event Problem Codes (Refer to coding manual) | Stathed | |
| Age of Device | | |
| Pailent | Results | |
| Device | Ocndusians - | <b>-</b> |
| Code | | . Vince of Marine |
| 11. Report Sent to FDA? | | 8. Visage of Bevioa Index Use of Device |
| Yes Hossital Obgostic Facility | ☐ Recall ☐ Notification | Repse |
| No (mo/day/yr) Hame Ambelstory | Repair inspection | Ustrons |
| 13. Report Sent to Manufacturer? Murping Home Surgical Facility | Replace Pallent Monitoring | S. If action reported to FDA under |
| Outputient Tresument Facility | Relabeting Matification/ | 21 USC \$80(f), list correction/<br>removal reporting number. |
| No (morbsy)t/) Crest | Oiber: | temeral industrial transman. |
| (Specify) | | |
| *4. Manufacturer Hame/Address | 13 Addžionai Manufacturer Narrative | and for 11 Corrected Data |
| G. ALL MANUFACTURIERS 5. Ganisol Office - Name/Address (and Manufacturing Sile 2. Phone Number | _ | |
| for Devises) | | |
| 3. Report Source<br>(Onect all that apply) | | |
| Foreign | | |
| ☐ Ziudy | | |
| ☐ Consumer | | |
| Health Professional | | |
| ☐ User Facility | | |
| II. Date Received by | | |
| Representative | | ; |
| Obstanter ND ± Distanter | | |
| PLA# | | |
| Pre4938 Yes | | |
| (These of Hepton OTC Tyes | | |
| Product Product S. Adverso Event Tormic) | | |
| S. Adversed Events and to the control of the contro | | |
| ☐ Indiai ☐ Follow to # | | |
| 5. Manufacturer Report Number | | |
| The public reporting burden for this policities of information has been estimated to exerage one | Department of Health and Homan Services | OMB Blatement:<br>'An agency may not conduct or position, |
| hour may recovere including the time for reviewing instructions, realizability safating data | Food and Drug Administration | - 1855 · 5 · 5 · 6 · 6 · 6 · 19 · 76 · 6 · 19 · 10 · 10 · 10 · 10 · 10 · 10 · 10 |
| courses, galheding and maintaining the data necest, and completing and texteating the colection of information. Send comments regarding this builden estimate or any other aspect of this collection of information, including suggestions for recording this Exteen to: | Medikiston; HPD-418<br>6603 Fishers Lane<br>Rockylle, MD 36657 | To, a collection of information unless to cisplays a currently valid OMB contractionable." |

Protocol: FVF3817s Final

34

#### APPENDIX D

## Analysis of Similar Events Template for IND Safety Reports

## **IND Safety Report**

## **Case Summary**

This section will be initiated by a research coordinator and may be modified by principal investigators if necessary. The case summary should describe the reported AE in detail, including a description of what happened and a summary of all relevant clinical information (e.g. medical status prior to the event, signs, symptoms, diagnoses, clinical course, treatment, outcome, etc.) The IND safety report should not identify the subject ID #, reporting investigator, or the site as this information may compromise the study blind.

#### **PREVIOUS REPORTS**

The information for this section comes from Principal Investigator and the search of similar events. This section should be written by the responsible principal investigator.

| <ul> <li>Select one of the following t</li> </ul> | wo statements after reviewing the s | earch of similar events results. |
|---|---|---|
| Under IND(insert INI submitted: | D#), the following IND safety reports | of similar AEs have been previously |
| MCN | Reported Event | Submission Date |
| | Or | |
| Under IND (insert IN previously | D#), no IND safety reports of similar | AEs have been submitted |
| pervious serious reports of the<br>product at the time of the repor-<br>made by an Independent Mon-<br>what similar events to summa<br>report generated by Clinical D | same/similar event that were consi | after reviewing the similar events is particularly worrisome (e.g., a |
| Assessment of Relationship | | |
| After evaluation the new case PI selects one of the following alternative conclusion | report and reviewing any relevant p<br>boilerplate conclusion statements, i | revious reports of similar events, the if applicable. The PI may also craft an |
| possibility of a cause-and-effe | data, Rush University Medical Cente<br>ct relationship between administrations<br>ce of( insert AE). | er believes there is a reasonable on of(insert study |
| Additional information on risk | factors and/or treatment of the AE m | nay be provided if warranted |

Protecol: FVF3817s Final 28DEC06

Or

| Based on review of available data, Rush University Medical Center does not believe that there is a reasonable possibility of a cause-and-effect relationship between administration of(insert study drug name) and the occurrence of(insert AE) |
|---|
| Explain if warranted. Do not speculate. |
| Or |
| Based on review of available data, Rush University Medical Center cannot establish or exclude the possibility of a cause-and-effect relationship between administration of(insert study drug name) and the occurrence of(insert AE) |
| Explain if warranted Do not speculate |
| After review of the clinical details and investigator's comments pertaining to this AE, and based on experience to date, Rush University Medical Center does not believe that changes to the conduct of this clinical trial are warranted This statement can be modified if changes to the conduct of the clinical trial are made |

Protocol: FVF3817s Final

36